CLINICAL TRIAL: NCT03426527
Title: Levobupivacaine Versus Levobupivacaine - Dexmedetomidine for Ultrasound Guided Bilateral Superficial Cervical Plexus Block for Upper Tracheal Resection and Reconstruction Surgery Under General Anesthesia
Brief Title: Dexmedetomidine for Bilateral Superficial Cervical Plexus Block for Reconstructive Tracheal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R/17.09.19
Record Dates: First submitted 2018-01-31; First posted 2018-02-08 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Tracheal Reconstruction
MeSH Terms: interventions — Levobupivacaine; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levobupivacaine (Placebo Comparator): Patients will receive bilateral superficial cervical plexus block using levobupivacaine General anesthesia
  Interventions: Drug: Levobupivacaine; Other: General Anaesthesia
- Levobupivacaine-Dexmedetomidine (Active Comparator): Patients will receive bilateral superficial cervical plexus block using levobupivacaine-dexmedetomidine General anesthesia
  Interventions: Drug: Levobupivacaine-Dexmedetomidine; Other: General Anaesthesia

INTERVENTIONS:
Drug: Levobupivacaine — Following induction of anaesthesia, patients will receive ultrasound guided bilateral superficial cervical plexus block with levobupivacaine
  Arms: Levobupivacaine
Drug: Levobupivacaine-Dexmedetomidine — Following induction of anaesthesia, patients will receive ultrasound guided bilateral superficial cervical plexus block with levobupivacaine in conjunction with dexmedetomidine
  Arms: Levobupivacaine-Dexmedetomidine
Other: General Anaesthesia — Using propofol, fentanyl and atracurium

SUMMARY:
Tracheal resection and reconstruction (TRR) is the treatment of choice for most patients with tracheal stenosis or tracheal tumors .The post intubation tracheal stenosis is the common indication for (TRR).The immediate postoperative period can be anxiety provoking for some reasons such as requirement to maintain a flexed neck, oxygen mask, and surgical pain which inadequately treated.

Bilateral superficial cervical plexus block (BSCPB) is a popular regional anesthesia technique for its feasibility and efficacy. The use of regional anesthesia in combination with general anesthesia may lighten the level of general anesthesia required , provide prolonged postoperative analgesia and reduce the requirements for opioid analgesics

Dexmedetomidine is a highly selective α2 agonist with high affinity for α2 adrenergic receptors and less α1 effects, which is responsible for the hypnotic and analgesic effects. Previous trials demonstrated that perineural dexmedetomidine in combination with bupivacaine enhanced sensory and motor block ,without neurotoxicity ,in both experimental and clinical studies.

Levobupivacaine, is "S"-enantiomer of bupivacaine, has strongly emerged as a safer alternative for regional anesthesia than bupivacaine . Levobupivacaine has been found to be equally efficacious as bupivacaine, but with a superior pharmacokinetic profile.

Clinically, levobupivacaine has been observed to be well tolerated in regional anesthesia techniques both after bolus administration and continuous post-operative infusion.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the intra- and postoperative efficacy of levobupivacaine versus levobupivacaine - dexmedetomidine for superficial cervical plexus block for upper tracheal resection and reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I or II.

Exclusion Criteria:

* History of allergy to the drugs used
* Coagulation disorders
* Pregnancy
* Postpartum period.
* Lactating females
* Local sepsis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Cumulative postoperative opioid consumption | For 24 hours after surgery
  Total postoperative opioid consumption

SECONDARY OUTCOMES:
Systolic blood pressure | Before and for 6 hours after start of anaesthesia
  Perioperative changes in systolic blood pressure
Diastolic blood pressure | Before and for 6 hours after start of anaesthesia
  Perioperative changes in diastolic blood pressure
Heart rate | Before and for 6 hours after start of anaesthesia
  Perioperative changes in heart rate
Peripheral oxygen saturation | Before and for 6 hours after start of anaesthesia
  Perioperative changes in peripheral oxygen saturation
End-tidal carbon dioxide tension | Before and for 6 hours after start of anaesthesia
  Perioperative changes in end-tidal carbon dioxide tension
Time for first analgesic request of analgesia following extubation | For 24 hours after surgery
  Time to receiving the rescue analgesic following surgery
Pain scores | For 24 hours after surgery
  Using visual analogue score (it is 100 mm unmarked line in which 0 = no pain and 100 = worst pain),score >30 mm needs rescue analgesics
Cortisol serum level | before induction of anaesthesia , one hour after the block then one hour after recovery
  Perioperative changes in cortisol level

CONTACTS AND LOCATIONS:
Overall Officials: Salwa MS Hayes, MD, Study Chair — Assistant Professor, MD anesthesia Department, Faculty of Medicine, Mansoura University, Egypt.
Locations (1):
- Mansoura University, Central Hospital, Oto-Rhino-Laryngology anesthesia Unit, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided